CLINICAL TRIAL: NCT06599853
Title: Evaluation of the Effect of Fever Education Given to Parents of Children Presenting to the Emergency Department With Fever on Parental Anxiety Level and Fever Management
Brief Title: Fever Education Given to Parents of Children Presenting to the Emergency Department With Fever
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merve YETİMOĞLU (Other)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Sponsor-Investigator, Merve YETİMOĞLU, Nursing, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KaradenizTU-SBF-MY-01
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fever
Keywords: Emergency; Fever; Parents; Education; Child; Anxiety
MeSH Terms: conditions — Fever; Emergencies; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The research was planned as a randomized controlled study with experimental and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group to be trained (Experimental): Parents in the experimental group were randomly assigned. Parents in the experimental group will be trained with parent fever management training material via home visits. Repeated measurements will be made one month after the training and at 3 months. Parent fever management training material was created by the researcher according to the literature. Opinions of experts in the field were obtained for the suitability of the training booklet.
  Interventions: Other: Fever Education
- Control group (No Intervention): No intervention will be made to the control group. Only measurements will be made on parallel dates with the experimental group.

INTERVENTIONS:
Other: Fever Education — Another aspect of this research that is different from other studies is that a retention test will be applied to the participants after the pre-test and post-test, and the long-term effect of the training given will be examined. In this direction, it is aimed to reduce the inappropriate use of emergency services, the use of unnecessary tests and the increasing health system costs. It is aimed to prevent crowding in the emergency department by reducing the inappropriate use of emergency services.
  Other Names: It is planned to conduct a survey with the first post-test and a retention test 3 months after the training is given to the parents.
  Arms: Group to be trained

SUMMARY:
Fever is a common symptom of childhood, especially between the ages of one and five, and is the main reason for emergency room visits. These emergency room visits are due to parents incorrect information and practices regarding fever management. This situation causes an increase in parental anxiety and failure to provide fever management. In line with this information, this study was planned to evaluate the effects of education given to parents of children presenting to the emergency room with fever on parental anxiety level and fever management.

DETAILED DESCRIPTION:
Fever is a common symptom in childhood and is the main reason for emergency room visits. The rate of children applying to the emergency department due to fever in our country is quite high compared to the rest of the world. Parents misinformation and practices regarding fever increase parental anxiety levels and negatively affect fever management. Interventional studies aimed at reducing parents anxiety levels and ensuring fever management are quite limited. This research will evaluate the effect of fever education given to parents on their anxiety levels and fever management.

The research was planned as a randomized controlled study with experimental and control groups. The research will be carried out between April 2024 and April 2025. After the power analysis of the sample, a total of 80 people will be included in the sample, 40 in the experimental group and 40 in the control group. Parents in the experimental group will be given fever training, while parents in the control group will not receive any treatment. Data will be collected with Parent-Child Introductory Information Form, State Anxiety Scale, Parent Fever Management Scale, Visual Analogue Scale (VAS)- Satisfaction with Fever Education Practice Scale and Parent-Education Satisfaction Form Scale. The data will be pre-tested, post-tested 1 month after the training, and permanence tested 3 months after the training, and the research will be terminated. Generalised linear models analysis, robust ANOVA, independent samples t test, Mann Whitney U and chi-square analysis will be used in the evaluation of the data. Mean, s.deviation, median, minimum and maximum will be used for quantitative data and frequency and percentage will be used for categorical data.As a result of the research, it is expected that fever education given to parents will positively affect parental anxiety level and fever management.

ELIGIBILITY:
Inclusion Criteria:

* Having a child between the ages of 1-5
* Able to read, understand and have no problems speaking Turkish
* Having a green triage code in the emergency room triage application

Exclusion Criteria:

* Children diagnosed with or receiving treatment for chronic diseases
* Children with a history of febrile convulsions
* Children dependent on home mechanical ventilation
* Parents with psychiatric diagnoses will be excluded from the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | one months
  This form was prepared by the researcher in line with the literature. This form consists of three sections. The parent sociodemographic form, the child sociodemographic form and the form, which includes questions on parental fever-related knowledge and practices, consists of a total of 35 questions.
State/Trait Anxiety Inventory (SAI) | one months
  The scale was developed by Spielber and others in 1964 to determine anxiety levels. The Turkish validity and reliability of the scale was carried out by Öner and Le Compte in 1985. The scale provides information about what is felt at that moment and consists of 20 items in Likert type, scored from 1 to 4. 1 is not at all, 2 is a little, 3 is very much and 4 is completely agree, and the individual marks one of these. A value of 1 indicates high anxiety, while a value of 4 indicates low anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 in the SAI are reversed. When calculating the scale score, the total score of the reversed items is subtracted from the total of the correct statements and a fixed score of 50 is added to this number. The total score obtained from the scale varies between 20 and 80. As the score increases, it indicates that anxiety is high, and as the score decreases, it indicates that anxiety decreases.
Parental Fever Management Scale-Turkish Version (PFMS-TR) | one months
  The scale was developed by Walsh and Edwards in 2008 to assess parents' fever management practices. The Turkish validity and reliability of the scale was conducted by Cınar et al. in 2013. The scale consists of 8 items and is a Likert-type scale with items rated as "(1) never, (2) rarely, (3) sometimes, (4) often, (5) always". The lowest possible score for the scale is 8 and the highest is 40. A higher score indicates more fever management practices, and a lower score indicates less fever management practices. The Cronbach Alpha reliability coefficient of the scale is 0.75.

SECONDARY OUTCOMES:
State/Trait Anxiety Inventory (SAI) | three months
  The scale was developed by Spielber and others in 1964 to determine anxiety levels. The Turkish validity and reliability of the scale was carried out by Öner and Le Compte in 1985. The scale provides information about what is felt at that moment and consists of 20 items on a Likert-type scale scored from 1 to 4. 1 is not at all, 2 is a little, 3 is very much, and 4 is completely agree, and the individual marks one of these. A value of 1 indicates high anxiety, while a value of 4 indicates low anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 on the SAI are reversed. When calculating the scale score, the total score of the reversed items is subtracted from the total of the correct statements and a fixed score of 50 is added to this number. The total score obtained from the scale varies between 20 and 80. As the score increases, it indicates that anxiety is high, and as the score decreases, it indicates that anxiety decreases.
Visual Analog Scale (VAS) - Satisfaction Scale for Fire Education Application | three months
  The scale was developed by Hayes and Patterson in 1921 and is a scale used to measure some expressions with numbers. Two expressions to be evaluated on a straight line are at two extreme points. The line contains numbers from 1 to 10. The participant is asked to mark the point that describes his/her own situation. It was planned to measure satisfaction with the fire education application by taking the Visual Analog Scale as an example. I am not satisfied at one end of the line, and I am very satisfied at the other end, and the parent will be asked to evaluate his/her situation.
Parental Fever Management Scale-Turkish Version (PFMS-TR) | three months
  The scale was developed by Walsh and Edwards in 2008 to assess what parents do in fever management. The Turkish validity and reliability of the scale was carried out by Cınar et al. in 2013. The scale consists of 8 items and is a Likert-type scale where the items are graded as "(1) never, (2) rarely, (3) sometimes, (4) often, (5) always". The lowest possible score for the scale is 8 and the highest is 40. A higher score indicates that more fever management practices are being implemented, and a lower score indicates that fewer fever management practices are being implemented. The Cronbach Alpha reliability coefficient of the scale is 0.75.
Parental Fever Management Scale-Turkish Version (PFMS-TR) | two months
  The scale was developed by Walsh and Edwards in 2008 to assess what parents do in fever management. The Turkish validity and reliability of the scale was carried out by Cınar et al. in 2013. The scale consists of 8 items and is a Likert-type scale where the items are graded as "(1) never, (2) rarely, (3) sometimes, (4) often, (5) always". The lowest possible score for the scale is 8 and the highest is 40. A higher score indicates that more fever management practices are being implemented, and a lower score indicates that fewer fever management practices are being implemented. The Cronbach Alpha reliability coefficient of the scale is 0.75.
State/Trait Anxiety Inventory (SAI) | two months
  The scale was developed by Spielber et al. in 1964 to determine the level of anxiety. The Turkish validity and reliability of the scale was carried out by Öner and Le Compte in 1985. The scale provides information about what is felt at that moment and consists of 20 Likert-type items scored from 1 to 4. 1 is not at all, 2 is a little, 3 is very much and 4 is completely agree, and the individual marks one of these. A value of 1 indicates high anxiety, while a value of 4 indicates low anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 in the SAI are reversed. When calculating the scale score, the total score of the reversed items is subtracted from the total of the correct statements and a fixed score of 50 is added to this number. The total score obtained from the scale varies between 20 and 80. A higher score indicates that anxiety is high, and a lower score indicates that anxiety is decreasing.

CONTACTS AND LOCATIONS:
Overall Officials: Merve YETİMOĞLU, Nursing, Principal Investigator — Karadeniz Technical University
Locations (2):
- Turkey (Türkiye) (2):
  - Karadeniz Technical University Faculty of Medicine Pediatric Emergency Unit, Trabzon, Kanuni Campus
  - Karadeniz Technical University Faculty of Medicine Pediatric Emergency Unit, Trabzon

IPD SHARING:
Plan to Share IPD: No